CLINICAL TRIAL: NCT04850898
Title: A Phase 2a, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety and Treatment Efficacy of SAB-176 (a Quadrivalent Anti-seasonal Influenza Immunoglobulin Product) in an H1N1 Challenge Model in Healthy Adult Participants
Brief Title: Study of SAB-176 in Healthy Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Collaborators: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAB-176-201
Record Dates: First submitted 2021-04-06; First posted 2021-04-20 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Influenza A H1N1
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Intervention Model Description: Exploratory randomised, Phase 2a, double blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal Saline Placebo Control (Placebo Comparator): Placebo control dosed 1 time via intravenous infusion
  Interventions: Other: Placebo
- SAB-176 - 25mg/kg (Experimental): Investigational Medicinal Product dosed 1 time at 25 mg/kg on day 1 via intravenous infusion
  Interventions: Biological: SAB-176

INTERVENTIONS:
Biological: SAB-176 — Treatment of influenza
  Arms: SAB-176 - 25mg/kg
Other: Placebo — Placebo Control
  Arms: Normal Saline Placebo Control

SUMMARY:
Healthy adult participants will be challenged with the H1N1 Influenza virus and then treated with either SAB-176 or placebo.

DETAILED DESCRIPTION:
Up to 60 eligible participants will be randomized in a 1:1 ratio to receive either SAB-176 (up to 25 mg/kg dose) or placebo. Healthy adult participants will be pre-screened for serosuitability for Influenza A/California/2009 H1N1 challenge virus. Serosuitable participants who sign the study specific informed consent form (ICF) will be challenged with an intranasal administration of Influenza A/California/2009 H1N1 virus on Day 0. Participants will be given intravenous (IV) infusion of SAB-176 or placebo on Day 1. Participants will be held in quarantine until Day 8.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the investigator
2. Aged between 18 and 45 years on the day of signing the study specific ICF.
3. In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination, (including vital signs), ECG, and routine laboratory tests as determined by the investigator.
4. A documented medical history prior to enrollment.
5. The following criteria are applicable to female participants:

   * Females of childbearing potential must have a negative pregnancy test prior to enrollment.
   * Females of non-childbearing potential:

   A.) Post-menopausal females: defined as having a history of amenorrhea for >12 months with no alternative medical cause, and/or by follicle stimulating hormone (FSH) level >40mIU/mL, confirmed by laboratory.

   b.) Documented status as being surgically sterile (e.g. tubal ligation, hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
6. The following criteria apply to female and male participants:

   a.) Female participants of childbearing potential must use one form of highly effective contraception. Hormonal methods must be in place from at least 2 weeks prior to the first study visit. The contraception used must continue until 28 days after the date of dosing with Investigational Medicinal Product (IMP)> Highly effective contraception is as described below:

   -Established use of hormonal methods of contraception described below (for a minimum of 2 weeks prior to the first study visit). When hormonal methods of contraception are used, male partners are required to use a condom with a spermicide: i.) Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: Oral, Intravaginal, or Transdermal ii.) progestogen-only hormonal contraception associated with inhibition of ovulation: Oral, Injectable, or Implantable

   b.) Intrauterine device c.) Intrauterine hormone-releasing system d.) bilateral tubal ligation e.) Male sterilization (with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate) where the vasectomised male is the sole partner for that woman.

   f.) True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

   B.) Male participants must agree to the contraceptive requirements below at entry to quarantine and continuing until 28 days after the date of dosing with IMP:
   1. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the IMP.
   2. Male sterilization with the appropriate post vasectomy documentation of the absence of sperm in in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure).
   3. In addition, for female partners of childbearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female participants.
   4. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

   C.) In addition to the contraceptive requirements above, male participants must agree not to donate sperm following discharge from quarantine until 28 days after the date of dosing with IMP.
7. Serosuitable to the Challenge virus, as defined in the study Analytical Plan (AP).

Exclusion Criteria:

(Participants are excluded from the study if any of the following criteria apply)

1. History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.

2.

1. Any history or evidence of any other clinically significant or currently active systemic comorbidities including psychiatric disorders (includes participants with a history of depression and/or anxiety).
2. And/or other major disease that, in the opinion of the investigator, may put the participant at undue risk, or interfere with a participant completing the stud and necessary investigations.

   The following conditions apply:
   * Participants with clinically mild atopic eczema/atopic dermatitis and clinically mild psoriasis may be included at the Investigator's discretion (e.g., if small amounts of regular topical steroids are used, no eczema in cubital fossa; moderate to large amounts of daily dermal corticosteroids is an exclusion).
   * Rhinitis (including hay fever) which is clinically active or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine will be excluded. Participants with a history of currently inactive rhinitis (within the last 30 days) or mild rhinitis may be included at the PI's discretion.
   * Participants with a physician diagnosed underactive thyroid who have been controlled on treatment for at least 6 months with evidence of a normal thyroid function test can be included at the discretion of the PI.
   * Any concurrent serious illness including history of malignancy that may interfere with the aims of the study or a participant completing the study. Basal cell carcinoma within 5 years of initial diagnosis or with evidence of recurrence is also an exclusion.
   * Participants with a history of psychiatric illness including depression and/or anxiety of any severity within the last 2 years can be included if the Patient Health Questionnaire (PHQ-9) and / or the Generalised Anxiety Disorder Questionnaire (GAD-7) is less than or equal to 4. Participants with a PHQ-9 or GAD-7 score of between 5 and 9 may be included following consultation with a Senior Physician (Clinical Lead for Screening) who may advise further consultation with the PI.
   * Participants reporting physician diagnosed migraine can be included provided there are no associated neurological symptoms such as hemiplegia or visual loss. Cluster headache/migraine or prophylactic treatment for migraine is an exclusion.
   * Participants with physician diagnosed mild irritable bowel syndrome not requiring regular treatment can be included at the discretion of the PI.

     3. Participants who have smoked ≥10 pack years at any time (10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years).

     4. A total body weight ≤50 kg or body mass index (BMI) ≤18 kg/m2 or ≥35 kg/m2.

     5. Females who: a) Are breastfeeding, or b) Have been pregnant within 6 months prior to the study.

     6. History of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.

     7. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
     1. Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and in particular any of the nasal assessments or viral challenge, (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month will be excluded).
     2. Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalised due to epistaxis on any previous occasion.
     3. Any nasal or sinus surgery within 3 months of the first study visit.

        PRIOR or CONCOMITANT MEDICATIONS AND ASSESSMENTS

        9.

     <!-- -->

     1. Evidence of vaccinations within the 4 weeks prior to the planned date of viral challenge, unless medically necessary (e.g., during an outbreak or pandemic situation) and at the PI's discretion.
     2. Intention to receive any vaccination(s) before the day of Follow-up visit. (NB. No travel restrictions will apply after the Day 28 Follow-up visit).
     3. Receipt of influenza vaccine in the last 6 months prior to the planned date of viral challenge.

        10. Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior to the planned date of viral challenge or planned during the 3 months after the final visit.

        11.

     <!-- -->

     1. Receipt of any investigational drug within 3 months prior to the planned date of viral challenge.
     2. Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge.
     3. Prior inoculation with a virus from the same virus-family as the Challenge virus.
     4. Prior participation in another Human Viral Challenge (HVC) study with a respiratory virus in the preceding 3 months, taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.
     5. Receipt of Polyclonal Antibodies (pAbs) or biologic within the previous 12 months prior to the planned date of viral challenge.

        12.

     a) Confirmed positive test for drugs of abuse and cotinine on first study visit. One repeat test allowed at PI discretion.

     b) History or presence of alcohol addiction, or excessive use of alcohol (weekly intake in excess of 28 units alcohol; 1 unit being a half glass of beer, a small glass of wine or a measure of spirits), or excessive consumption of xanthine containing substances (e.g., daily intake in excess of 5 cups of caffeinated drinks e.g., coffee, tea, cola).

     13. A forced expiratory volume in 1 second (FEV1) <80%.

     14. Positive HIV, active hepatitis A, B, or C test.

     15. Those employed or immediate relatives of those employed at hVIVO or the Sponsor.

     16. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Parker, Principal Investigator — hVIVO Services Limited
Locations (1):
- Queen Mary BioEnterprises Innovation Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 healthy adult participants were randomised and inoculated with the challenge virus of which 30 participants were treated with SAB-176 and 30 participants with placebo. Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
Pre-assignment Details: Two participants (1 in each treatment group) were inoculated with challenge virus but were not treated with Investigational Medicinal Product (IMP). In total, 60 participants were treated (30 with SAB-176 and 30 with placebo).
Period: Overall Study
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Started | 31 | 31
Completed | 30 | 30
Not Completed | 1 | 1
Not completed — Inoculated with challenge virus but were not treated with IMP | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants] — Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 29 | 30 | 59
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
  years | 24.5 [20 to 42] | 23 [18 to 45] | 23.5 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
  Participants
    Female | 8 | 10 | 18
    Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
  Participants
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 30 | 29 | 59
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants that were inoculated with challenge virus were not treated with investigational medicinal product (IMP) (1 in each treatment group) and were not included in the intent-to-treat (ITT) and safety analysis sets (and in the per protocol [PP], ITT-infected [ITT-I] or ITT-I sensitivity [ITT-Is] analysis sets).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 3 | 6
    White | 22 | 20 | 42
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Viral Load by Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR) of SAB-176 When Compared to Placebo
Description: Area under the viral load-time curve (VL-AUC) of Influenza A/California/2009 H1N1 virus, as determined by Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR) on nasal samples.
Time Frame: 28 Days
Population: All participants randomly assigned to study intervention who received the study intervention (ITT analysis set participants) who had no major protocol deviation likely to impact the efficacy evaluation, and who completed the quarantine period up to the final day of quarantine (Day 8) Participant 542996 was excluded from the PP analysis set due to a major protocol deviation prior to unblinding of treatment group assignment and primary and secondary endpoints were known.
Measure: Mean (Standard Deviation); unit: Log10 copies*hour/mL
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Log10 copies*hour/mL | 273.05 (337.247) | 91.98 (166.034)

2. Secondary Outcome: Evaluate Peak Viral Load Quantified by qRT-PCR.
Description: Peak viral load as defined by the maximum viral load determined by quantifiable qRT-PCR measurements to evaluate the effect of SAB-176 in reducing viral loads in qRT-PCR due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Log10 copies/mL | 3.8196 (3.73236) | 2.5440 (3.37243)

3. Secondary Outcome: Evaluate Duration of Influenza Quantified by qRT-PCR.
Description: Duration in hours of Influenza quantifiable qRT-PCR measurements to evaluate the effect of SAB-176 in reducing the duration of Influenza in qRT-PCR due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
hours | 1.3097 (1.90894) | 0.5503 (1.24432)

4. Secondary Outcome: Evaluate Peak Viral Load Determined by Cell Culture.
Description: Peak viral load as defined by the maximum viral load determined by quantifiable cell culture to evaluate the effect of SAB-176 in reducing viral loads in cell culture due to Influenza A/California/2009 H1N1 virus, compared to placebo.
Time Frame: 28 Days
Population: Participant 542996 was excluded from the PP analysis set due to a major protocol deviation prior to unblinding of treatment group assignment and primary and secondary endpoints were known.
Measure: Mean (Standard Deviation); unit: Log10 TCID 50/ml
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Log10 TCID 50/ml | 1.3097 (1.90894) | 0.5503 (1.24432)

5. Secondary Outcome: Evaluate Peak Viral Load Area Under the Curve Determined by Cell Culture.
Description: VL-AUC of Influenza A/California/2009 H1N1 virus as determined by cell culture to evaluate the effect of SB-176 in reducing viral loads in cell culture due to Influenza A/California/2009 H1N1 virus, compared to placebo.
Time Frame: 28 Days
Population: as for outcome 4
Measure: Mean (90% Confidence Interval); unit: hours * Log10 TCID 50/mL
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
hours * Log10 TCID 50/mL | 67.97 [33.55 to 102.40] | 7.99 [1.56 to 14.42]

6. Secondary Outcome: Duration of Influenza Using Peak Viral Load Determined by Cell Culture.
Description: Duration measured in hours of influenza quantifiable by cell culture measurement to evaluate the effect of SB-176 in reducing viral loads in cell culture due to Influenza A/California/2009 H1N1 virus, compared to placebo.
Time Frame: 28 Days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
hours | 1.3097 (1.90894) | 0.5503 (1.24432)

7. Secondary Outcome: TSS-AUC (Area Under the Curve Over Time of Total Clinical Symptoms Score) Measured by Graded Symptom Scoring System to Evaluate the Effect of SAB-176 in Reducing Symptoms Due to Influenza A/California/2009 H1N1 Virus Compared to Placebo.
Description: Using the hVIVO Symptom Diary Card, participants grade 11 distinct cold symptoms on a scale of 0-3 (Grade 0: No symptoms; Grade 1: just noticeable; Grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; Grade 3: Quite bothersome most or all the time, and it stops me participating in activities) and Shortness of Breath and Wheeze have a scale of 0-4 with 0-3 being the same and grade 4 being symptoms at rest. Additional to symptom card, a Visual Analogue Scale dairy card using a 0mm to 100mm scale, with the same 13 symptoms with 0mm being no symptoms. Total summed grading scale is 0 to 1341. Lower scores represent a better outcome.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total Symptom Score Scale-points*hour
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Total Symptom Score Scale-points*hour | 166.52 (282.313) | 51.06 (74.559)

8. Secondary Outcome: Peak Symptom Diary Card Score
Description: Peak symptom diary card score: peak total clinical symptoms (TSS) as measured by graded symptom scoring system to evaluate the effect of SAB-176 in reducing symptoms due to Influenza A/California/2009 H1N1 virus compared to placebo.
  Using the hVIVO Symptom Diary Card, participants grade 11 distinct cold symptoms on a scale of 0-3 (Grade 0: No symptoms; Grade 1: just noticeable; Grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; Grade 3: Quite bothersome most or all the time, and it stops me participating in activities) and Shortness of Breath and Wheeze have a scale of 0-4 with 0-3 being the same and grade 4 being symptoms at rest. Additional to symptom card, a Visual Analogue Scale dairy card using a 0mm to 100mm scale, with the same 13 symptoms with 0mm being no symptoms. Total summed grading scale is 0 to 1341. Lower scores represent a better outcome.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
score on a scale | 3.7 (4.79) | 1.8 (2.21)

9. Secondary Outcome: Peak Daily Symptom Score
Description: Peak symptom diary card score: The individual maximum daily sum of symptom score; peak TSS as measured by graded symptom scoring system to evaluate the effect of SAB-176 in reducing symptoms due to Influenza A/California/2009 H1N1 virus compared to placebo.
  Using the hVIVO Symptom Diary Card, participants grade 11 distinct cold symptoms on a scale of 0-3 (Grade 0: No symptoms; Grade 1: just noticeable; Grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; Grade 3: Quite bothersome most or all the time, and it stops me participating in activities) and Shortness of Breath and Wheeze have a scale of 0-4 with 0-3 being the same and grade 4 being symptoms at rest. Additional to symptom card, a Visual Analogue Scale dairy card using a 0mm to 100mm scale, with the same 13 symptoms with 0mm being no symptoms. Total summed grading scale is 0 to 1341. Lower scores represent a better outcome.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
score on a scale | 8.3 (11.24) | 3.6 (5.31)

10. Secondary Outcome: Percent of Participants With Grade 2 or Higher Symptoms.
Description: Number (percent) of participants with Grade 2 or higher symptoms to evaluate the effect of SAB-176 in reducing symptoms due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
percentage of participants | 30 [18.37 to 44.94] | 20.7 [11.10 to 35.29]

11. Secondary Outcome: RT-PCR Confirmed Symptomatic Influenza Infection.
Description: RT-PCR-confirmed influenza infection (any 2 quantifiable [≥ lower limit of quantification {LLOQ}] qRT-PCR measurements reported) over 4 consecutive scheduled timepoints, from morning of Day 2 up to Day 8 (discharge from quarantine) AND clinical symptoms (grade 2 or more symptoms) between Day 2 and quarantine discharge.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Participants | 15 | 9

12. Secondary Outcome: Culture Lab-confirmed Reduction of Symptomatic Influenza Infection.
Description: Culture lab-confirmed reduction of symptomatic influenza infection defined as: lab-confirmed culturable influenza infection and clinical symptoms to evaluate the effect of SAB-176 in reducing the incidence of symptomatic infection due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: RT-PCR-confirmed influenza infection (any 2 quantifiable [≥lower limit of quantification {LLOQ}] qRT-PCR measurements reported) over 4 consecutive scheduled timepoints, from morning of Day 2 up to Day 8 (discharge from quarantine) AND clinical symptoms (grade 2 or more symptoms) between Day 2 and quarantine discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Participants | 6 | 2

13. Secondary Outcome: Total Number of Participants That Any Adverse Event (AE) Was Reported for Which Occurred Across All Participants From IV Infusion up to Day 28 Follow-up.
Description: Total number of participants that any adverse events (AEs) that occurred across all participants was reported; Captured from IV infusion up to Day 28 follow-up to evaluate the safety of SAB-176 when compared to placebo.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 30
Participants | 16 | 18

14. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs) From IV Infusion up to Day 28 Follow up.
Description: Total number, by occurrence, of serious adverse events (SAEs) from IV infusion up to Day 28 follow up to evaluate the safety of SAB-176 when compared to placebo.
Time Frame: 28 Days
Population: All participants who signed an Informed Consent. Two participants (1 in each treatment group) were inoculated with challenge virus but were not treated with IMP.
Measure: Number; unit: SAE occurrence
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 31 | 31
SAE occurrence | 0 | 0

15. Other Pre Specified Outcome: Number of Participants With Upper Respiratory Tract Illness.
Description: Evaluate number of participants with upper respiratory tract illness to determine the effect of SAB-176 in reducing the incidence of influenza illness due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Participants | 6 | 5

16. Other Pre Specified Outcome: Number of Participants With Lower Respiratory Tract Illness.
Description: Evaluate number of participants with lower respiratory tract illness to determine the effect of SAB-176 in reducing the incidence of influenza illness due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
participants | 3 | 0

17. Other Pre Specified Outcome: Number of Participants With Systemic Illness.
Description: Evaluate number of participants with systemic illness to determine the effect of SAB-176 in reducing the incidence of influenza illness due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Participants | 4 | 2

18. Other Pre Specified Outcome: Number of Participants With Mild to Moderate Symptoms.
Description: Evaluate number of participants with mild to moderate symptoms to determine the effect of SAB-176 in reducing the incidence of influenza illness due to Influenza A/California/2009 H1N1 virus compared to placebo.
Time Frame: 28 Days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
percentage of participants | 30 [18.37 to 44.94] | 20.7 [11.10 to 35.29]

19. Other Pre Specified Outcome: Influenza Viral Infection Rates in Upper Respiratory Samples by qRT-PCR
Description: Influenza viral infection rates in upper respiratory samples by qRT-PCR to explore the effect of SAB-176 in reducing the incidence of infection due to Influenza A/California H1N1 Virus.
Time Frame: 28 Days
Population: Participant 542996 was excluded from the PP analysis set due to a major protocol deviation prior to unblinding of treatment group assignment and primary and secondary endpoints were known. RT-PCR-confirmed influenza infection (any 2 quantifiable [≥lower limit of quantification {LLOQ}] qRT-PCR measurements reported) over 4 consecutive scheduled timepoints, from morning of Day 2 up Day 8 (discharge from quarantine) AND clinical symptoms (grade 2 or more symptoms) between Day 2 and discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline Placebo Control | SAB-176 - 25mg/kg
Number analyzed (Participants) | 30 | 29
Participants | 8 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the signing of the Informed Consent Form on Day -56 to the last follow up on Day 28 (a duration of approximately 12 weeks).
Description: The PI is responsible for ensuring that all AE/SAEs, and pregnancies are identified, evaluated, recorded, and reported. Ensures that the medical mgt of AEs, SAEs and, pregnancy symptoms is provided by competent Investigator. The definitions of an AE or SAE, as well as the method of recording, evaluating, and assessing causality of AE/SAE and the procedures for completing and transmitting AE, SAE, and other reportable safety event reports can be found in Appendix 3 of the protocol.
Groups:
- Normal Saline Placebo Control: Participants randomized to the control (placebo) infusion will receive normal (0.9%) saline in approximately the same volume as they would have received if randomized to the active arm.
- SAB-176: SAB-176 is diluted in normal (0.9%) sterile saline under aseptic conditions. The diluted product is intended for administration by the IV route. The dose of IMP will be calculated. The pharmacy will prepare a bag containing the dose of SAB-176 plus as much normal (0.9%) saline as is needed to reach the concentrations for the study.
Arm/Group | Normal Saline Placebo Control | SAB-176
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04850898/Prot_SAP_000.pdf